CLINICAL TRIAL: NCT01948115
Title: Prospective Randomized Controlled Trial to Evaluate the Efficacy and Safety of an Equimolar Mixture of Oxygen and Nitrous Oxide in External Cephalic Version (ECV) in Singleton Pregnancy in Breech Presentation at Term
Brief Title: Evaluation of the Efficacy and Safety of an Equimolar Mixture of Oxygen and Nitrous Oxide in External Cephalic Version (ECV)
Acronym: MEOREV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC13_0254
Record Dates: First submitted 2013-09-15; First posted 2013-09-23 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-11

CONDITIONS: Breech Presentation in Pregnancy
Keywords: Breech presentation; equimolar mixture of oxygen and nitrous oxide; external cephalic version
MeSH Terms: conditions — Breech Presentation | interventions — Nitrous Oxide; Air

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical air (Placebo Comparator)
  Interventions: Drug: equimolar mixture of oxygen and nitrous oxide or medical air
- equimolar mixture of oxygen and nitrous oxide (Experimental)
  Interventions: Drug: equimolar mixture of oxygen and nitrous oxide or medical air

INTERVENTIONS:
Drug: equimolar mixture of oxygen and nitrous oxide or medical air — We need to include 150 patients for a period of 2 years. Patients will be randomized: 75 patients in each arm: 75 patients in group "placebo" (medical air), 75 patients in group "treatment" (equimolar mixture of oxygen and nitrous oxide).
  Patients will be single-blind. The ECV be started at least 3 minutes after the start of administration. The maximum time of administration of the gas will be 15 minutes. Just after ECV, we compare success rate of intervention.

SUMMARY:
The variety of breech presentation at term is about 3-4% of all births. Our study aims to assess the value of using an equimolar mixture of oxygen and nitrous oxide. Indeed, in some patients algic or relaxed, the success rate seems more important.

It's a single blind prospective randomized controlled study, comparing success rate of ECV after an equimolar mixture of oxygen and nitrous oxide or placebo (medical air).

We need to include 150 patients (75 in each arm), for a period of 2 years. After ECV, we will give the patient a satisfaction questionnaire. We compare the success rate of ECV as primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* pregnancy at term (≥36 weeks)
* singleton foetus in breech or transverse presentation
* acceptance of ECV
* signature of informed consent

Exclusion Criteria:

* contraindications of ECV: placenta praevia, obstacle praevia, multiple pregnancy, foetal death, foetal heart rhythm disorder, lack of amniotic fluid, HIV-positive patient
* contraindications of equimolar mixture of oxygen and nitrous oxide : patient who require pure oxygen ventilation, disorders of consciousness that impede the cooperation of the patient, pneumothorax, pulmonary embolism, ocular surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of women with success after ECV | 20 minutes
  Success rate just after ECV between the two groups (equimolar mixture of oxygen and nitrous oxide group, and medical air group) with ultrasound.

SECONDARY OUTCOMES:
Pain during ECV | 20 minutes
  Just after ECV:
  pain during ECV with Visual Analogue Scale
Frequency of nausea/vomiting | 1 hour
  Just after ECV:
  Frequency of nausea / vomiting between the two groups
Number of interrupted procedures | 20 minutes
  Just after ECV:
  number of interrupted procedures due to pain
Number of cephalic presentation at birth | 2 month
  At birth:
  rate of cephalic presentation between the two groups
Number of cesarean at birth | 2 month
  At birth:
  cesarean rate between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Julie ESBELIN, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Derived] Dochez V, Esbelin J, Misbert E, Arthuis C, Drouard A, Badon V, Fenet O, Thubert T, Winer N. Effectiveness of nitrous oxide in external cephalic version on success rate: A randomized controlled trial. Acta Obstet Gynecol Scand. 2020 Mar;99(3):391-398. doi: 10.1111/aogs.13753. Epub 2019 Nov 18. PMID 31630398